CLINICAL TRIAL: NCT01122875
Title: An Open-Label, Multicenter, Phase I Trial of the Safety and Pharmacokinetics of Escalating Doses of MFGR1877S in Patients With Relapsed or Refractory t(4;14)-Positive Multiple Myeloma
Brief Title: A Study of the Safety and Pharmacokinetics of MFGR1877S in Patients With Relapsed or Refractory t(4;14)-Positive Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MFG4809g; GO01331 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — vofatamab

ARMS (1):
- A (Experimental)
  Interventions: Drug: MFGR1877S

INTERVENTIONS:
Drug: MFGR1877S — Intravenous repeating dose

SUMMARY:
This is a multicenter, open-label, dose-escalation study of MFGR1877S in patients with relapsed or refractory t(4;14)-positive multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0, 1, or 2
* Life expectancy of at least 12 weeks
* Histologic documentation of previously treated t(4;14)-positive multiple myeloma for which no effective standard therapy exists

Exclusion Criteria:

* Prior use of any monoclonal antibody before study treatment
* Treatment with radiotherapy, thalidomide, lenalidomide, bortezomib, any chemotherapeutic agent, or treatment with any other investigational anti-cancer agent within 4 weeks of study treatment
* Completion of autologous stem cell transplant within 6 months prior to study treatment
* Prior allogeneic stem cell transplant
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
* Evidence of significant, uncontrolled concomitant diseases, including significant cardiovascular disease or pulmonary disease
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection at screening or any recent major episode of infection requiring treatment with IV antibiotics or hospitalization prior to study treatment
* Recent major surgery (prior to study treatment), other than for diagnosis
* Presence of positive test results for Hepatitis B or Hepatitis C
* Known history of HIV seropositive status
* Women who are pregnant or lactating
* Childbearing potential without agreement to use effective form of contraception for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of dose-limiting toxicities (DLTs) | Throughout study or until early study discontinuation

SECONDARY OUTCOMES:
Incidence, nature, and severity of adverse events | Throughout study or until early study discontinuation
Clinical activity of MFGR1877S (objective response, duration of response, and progression-free survival) | Throughout study or until early study discontinuation
Pharmacokinetic parameters of MFGR1877S (total exposure, maximum and minimum serum concentrations, clearance, volume of distribution) | Throughout study or until early study discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (12):
- United States (11):
  - Scottsdale, Arizona
  - Atlanta, Georgia
  - Chicago, Illinois
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Hackensack, New Jersey
  - New York, New York
  - Dallas, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
- Toronto, Ontario, Canada